CLINICAL TRIAL: NCT03334838
Title: Open-label, Randomized, Single-dose, Cross-over Study to Evaluate the Influence of Dietary Habits on the Pharmacokinetics, Safety, and Tolerability of a 120 mg Dose and to Assess the Relative Bioavailability of a 240 mg Dose of Nifurtimox Tablets Administered to Adult Male and Female Patients With Chagas' Disease
Brief Title: Study to Assess the Food Effect on the Pharmacokinetics of Nifurtimox Tablets in Chronic Chagas' Patients - Dietary Habits Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16006
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Chagas' Disease
Keywords: Food effect; Dose proportionality
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRP 1 - Assess relative bioavailability (4-way crossover) (Experimental): GROUP 1 (Treatments A, B, C, D) All treatments in Group 1 consisted of a dose of 120 mg nifurtimox (4 x 30 mg tablets).
  In Treatment A, dose administration was in a fasted state.
  For the other treatments, dose administration was in a fed state:
  Treatment B after a low-fat breakfast; Treatment C after a breakfast consisting of dairy products (yogurt+milk); and Treatment D after a high-calorie and high-fat breakfast.
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)
- GRP 2 - Assess relative bioavailability (2-way crossover) (Experimental): All subjects in Group 2 received a single dose of nifurtimox in each of the Treatments D and E.
  In Treatment D, subjects received 120 mg nifurtimox (4 x 30 mg tablets), and in Treatment E, subjects received 240 mg nifurtimox (8 x 30 mg tablets). Both treatments were administered in a fed state, after a high-calorie and high-fat breakfast.
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)

INTERVENTIONS:
Drug: Nifurtimox (Lampit, BAYA2502) — Oral Intake of 4 x 30 mg nufurtimox tablets for treatment A-D; Oral Intake of 8 x 30 mg nufurtimox tablets for treatment E.

SUMMARY:
This study evaluated the effect of food on the absorption of the drug as well as safety and tolerability in adults suffering from chronic Chagas' disease In addition pharmacokinetics of the drug following 120 and 240 mg single doses will be assessed

DETAILED DESCRIPTION:
Primary objective was to evaluate the effect of various food compositions on the PK of nifurtimox after a single oral dose (120 mg) administered under 3 types of fed conditions (low fat, dairy products, and high calorie and high fat), as well as fasted conditions, to assess relative bioavailability. It was chosen to allow a direct inter-study comparison of PK data obtained in previous studies.

A secondary objective of the study was to assess the relative bioavailability of 2 different dose levels of nifurtimox, given as a single oral dose, in a second group of patients.The second treatment group addressed a biopharmaceutical aspect for which no study data have been obtained to date. In order to assess the relationship between dose and exposure (linearity of PK), an analysis of the dose range of 120 mg to 240 mg was chosen to close the knowledge gap for this dose range.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be provided before any study-specific tests or procedures are performed.
* Male/female patient diagnosed with chronic Chagas' disease:

Previous diagnosis of acute or chronic Chagas' disease by a health clinic prior to screening for the study. The diagnosis of chronic Chagas' disease may be made by clinical findings, supported by antibody titers if available. If there is a known history of acute disease, it is preferable to have documentation of parasites on the blood smear, if available.

* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and 12 weeks after the last administration of study drug. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements. Acceptable methods of contraception include, but are not limited to: (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception. Subjects must agree to utilize two reliable and acceptable methods of contraception simultaneously.
* Women of childbearing potential with confirmed last menstrual period by anamnesis and negative serum pregnancy test (beta-human chorionic gonadotropin [βhCG]) at screening and negative urine pregnancy test (βhCG) at pre-dose of each treatment.
* Women of non-childbearing potential, such as surgically sterile women with either written documentation of surgical sterility or negative serum pregnancy test (βhCG) at screening and negative urine pregnancy test (βhCG) at pre-dose of each treatment.
* Male subjects who agree not to act as sperm donors for 12 weeks after last administration of study drug.
* Age: 18 to 45 years (inclusive) at screening.
* Body mass index (BMI): ≥18 and <29.9 kg/m².

Exclusion Criteria:

* Incompletely cured pre-existing diseases (except chronic Chagas' disease without active GI condition) for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study drugs will not be normal.
* Acute Chagas' disease. (During the acute phase, the parasite on a blood smear may be seen under a microscope. Different antibodies are present, depending on the course of the disease).
* Known hypersensitivity to the study drug (active substance or excipients of the preparations)
* Unstable or uncontrolled medical condition such as hypertension or diabetes, decompensated heart failure, GI conditions that would interfere with the absorption of the study drug (e.g. GI ulceration, peptic ulceration, GI bleeding, gastroesophageal reflux, or other GI disease affecting gastroesophageal junction), conditions that could potentially have an impact on drug metabolism or elimination (renal, hepatic such as known hepatic or biliary abnormalities), or any clinically relevant active infections in the opinion of the investigator within 4 weeks before the screening visit, e.g. clinically relevant history or presence of significant respiratory (e.g. interstitial lung disease), hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic (e.g. diabetes), and dermatological or connective tissue disease.
* Use of systemic or topical medicines or substances which oppose the study objectives (including clinical treatment with nifurtimox and benznidazole) or which might influence them within 4 weeks before the first study drug administration, e.g. an investigational drug, any drug altering GI motility and/or gastric pH (e.g. antacids, anticholinergic, para-sympatholytics), any drug known to induce liver enzymes (e.g. dexamethasone, barbiturates, St. John's Wort [hypericum perforatum]), any drug known to inhibit liver enzymes (e.g. ketoconazole, macrolides).
* Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over 120 msec or of the QT interval over 450 msec using Bazett's formula (QTcB). (Clinically stable subjects with Chagas'-related heart disease and pacemaker in place for >1 year and evaluated by a cardiologist ≤6 months before the first dose of study drug will not be excluded.)
* Systolic blood pressure <100 or >140 mmHg (after resting in supine position for a minimum of 3 minutes).
* Diastolic blood pressure <50 or >90 mmHg (after resting in supine position for a minimum of 3 minutes).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlast) of nifurtimox (evaluation of food effect) | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  Area under the drug-concentration vs. time curve of nifurtimox from time 0 to the last data point[AUC(0-tlast)]
Cmax of nifurtimox (evaluation of food effect) | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  Peak concentrations (Cmax) of the plasma concentration vs time profiles

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 8 weeks
  Clinical Laboratory Test, physical examinations, vital signs and 12 electrocardiograms ( ECG's) for safety and tolerability
AUC(0-tlast)/D of nifurtimox (evaluation of food effect) | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  AUC(0-tlast)/D: AUC(0-tlast) divided by dose
Cmax/D of nifurtimox (evaluation of food effect) | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  Cmax/D: Cmax divided by dose

CONTACTS AND LOCATIONS:
Locations (1):
- FP Clinical Pharma, Buenos Aires, Ciudad Auton. de Buenos Aires, Argentina

REFERENCES:
- [Derived] Stass H, Just S, Weimann B, Ince I, Willmann S, Feleder E, Freitas C, Yerino G, Munster U. Clinical investigation of the biopharmaceutical characteristics of nifurtimox tablets - Implications for quality control and application. Eur J Pharm Sci. 2021 Nov 1;166:105940. doi: 10.1016/j.ejps.2021.105940. Epub 2021 Jul 12. PMID 34265407